CLINICAL TRIAL: NCT01144156
Title: Small Bowel Mucosal Healing Induced by Adalimumab in Crohn's Disease Patients as Assessed by Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Dr Eyal Gal, Sherutei Briut Clalit
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Gal002
Record Dates: First submitted 2010-06-13; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Small bowel; Mucosal healing; Capsule endoscopy; Adalimumab; Small bowel Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Therapeutics; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Treatment with Adalimumab — All patients will receive SC adalimumab 160 mg at week 0, 80 mg at week 2 and 40 mg from week 4 every 2 weeks up to 12 weeks
  Other Names: Humira (Abbott Laboratories)

SUMMARY:
The study hypothesis is that adalimumab induces mucosal healing in the small bowel and that mucosal healing correlates with disease activity. 30 Patients with isolated active small bowel Crohn's disease which are candidates to receive anti-TNF treatment will be included in the study. All patients will undergo patency capsule examination and capsule endoscopy afterwards. Small bowel endoscopic disease severity will be assessed by the capsule endoscopy Crohn's disease activity index (CECDAI). The patients will receive Adalimumab (Humira)injections (160mg,80mg and 40mg every 2 weeks ) for 12 weeks. on week 14 a second capsule endoscopy will be performed and CECDAI calculated again. The patients clinical condition, CDAI,IBDQ and laboratory results including CRP, CBC and fecal calprotectin will be assessed on weeks o, 7 and 14 and results will be compared with the endoscopic score.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated small bowel Crohn's disease.
2. Age ≥18.
3. Active disease (CDAI≥220).

Exclusion Criteria:

1. Known fixed stricture in the small intestine.
2. Former small bowel obstruction or obstructive symptoms.
3. Patients expected to undergo small bowel surgery in the near future or had intestinal surgery in the previous 6 months.
4. Colonic disease (except ileocecal valve area).
5. Anti-TNF treatment in the last 3 months.
6. Sensitivity or lack of response to previous adalimumab treatment.
7. Current gastrointestinal infection.
8. History of malignant disease (except BCC of skin).
9. Congestive heart failure, severe renal or hepatic dysfunction.
10. Patients suffering from tuberculosis, hepatitis B or C.
11. Pregnancy or unwillingness to use contraception during study period.
12. Dysphagia or swallowing disorders
13. Gastroparesis or severe gastrointestinal motility dysfunction.
14. Patients with cardiac pacemaker or implanted cardioverter devices.
15. Unable to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)

PRIMARY OUTCOMES:
Complete mucosal healing | After 14 weeks of treatment
  Complete mucosal healing of active inflammatory lesions in the small intestine, as assessed by capsule endoscopy

SECONDARY OUTCOMES:
Partial mucosal healing | After 14 weeks of treatment
  Reduction of at least 50% in the Capsule Endoscopy Crohn's Disease Activity Index (CECDAI) after treatment.
Correlation with clinical activity | After 14 weeks of treatment
  Statistical correlation between CECDAI reduction and reduction in clinical (CDAI, IBDQ) and laboratory (CRP, calprotectin etc.) indices of disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] Gal E, Geller A, Fraser G, Levi Z, Niv Y. Assessment and validation of the new capsule endoscopy Crohn's disease activity index (CECDAI). Dig Dis Sci. 2008 Jul;53(7):1933-7. doi: 10.1007/s10620-007-0084-y. Epub 2007 Nov 22. PMID 18034304